CLINICAL TRIAL: NCT03234114
Title: Optimal Antithrombotic Therapy for Acute Coronary Syndrome Patients Concomitant With Atrial Fibrillation and Implanted With New-generation Drug-eluting Stent: OPTImal Management of Antithrombotic Agents (OPTIMA-3, 4)
Brief Title: Optimal Antithrombotic Therapy for ACS Patients Concomitant With AF and Implanted With New-generation DES (OPTIMA-3, 4)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Coronary Syndrome (ACS); Non-valvular Atrial Fibrillation (NVAF)
Keywords: new generation drug eluting stent (DES); antithrombotic therapy; randomized clinical trial (RCT)
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1-month TAT (Experimental): Randomized experimental group in the OPTIMA-3 substudy; Triple antithrombotic therapy (warfarin with targeted INR 2.0-3.0, clopidogrel 75 mg q.d. and aspirin 100 mg q.d.) for 1 month (30 days) then quit aspirin till 12 months after PCI
  Interventions: Drug: Triple antithrombotic therapy
- 6-month TAT (Experimental): Randomized control group in the OPTIMA-3 substudy; Triple antithrombotic therapy (warfarin with targeted INR 2.0-3.0, clopidogrel 75 mg q.d. and aspirin 100 mg q.d.) for 6 months (180 days）then quit aspirin till 12 months after PCI
  Interventions: Drug: Triple antithrombotic therapy
- 12-month DAT-1 (Experimental): Randomized experimental group in the OPTIMA-4 substudy; Dual antithrombotic therapy including dabigatran 110 mg b.i.d. with clopidogrel 75 mg q.d. for 12 months after PCI
  Interventions: Drug: Dual antithrombotc therapy-1
- 12-month DAT-2 (Experimental): Randomized control group in the OPTIMA-4 substudy; Dual antithrombotic therapy including dabigatran 110 mg b.i.d. with ticagrelor 90 mg b.i.d for 12 months after PCI
  Interventions: Drug: Dual antithrombotc therapy-2

INTERVENTIONS:
Drug: Triple antithrombotic therapy — Including warfarin with targeted INR 2.0-3.0 (Shanghai Xinyi pharma co., LTD, China), aspirin 100 mg q.d. (Bayer, Germany) and clopidogrel 75 mg q.d. (Sanofi, France)
  Other Names: TAT
  Arms: 1-month TAT; 6-month TAT
Drug: Dual antithrombotc therapy-1 — Including dabigatran 110 mg b.i.d. (Boehringer Ingelheim, Germany) plus clopidogrel 75 mg q.d. (Sanofi, France)
  Other Names: DAT-1
  Arms: 12-month DAT-1
Drug: Dual antithrombotc therapy-2 — Including dabigatran 110 mg b.i.d. (Boehringer Ingelheim, Germany) plus ticagrelor 90 mg b.i.d. (AstraZeneca, Britain)
  Other Names: DAT-2
  Arms: 12-month DAT-2

SUMMARY:
It is a multi-center randomized clinical trial (RCT) which will enroll 3746 patients with acute coronary syndrome (ACS) concomitant non-valvular atrial fibrillation (NVAF) and undergoing new generation drug eluting stent (DES) implantation at 70 centers nationwide in China and contains two sub-studies.

In the OPTIMA-3 sub-study, 2274 subjects who choose warfarin as anticoagulant will randomly receive triple antithrombotic therapy (warfarin with targeted INR 2.0-3.0, clopidogrel 75 mg od and aspirin 100 mg od) for 1 month or 6 months in a 1:1 ratio then quit aspirin till 12 months after percutaneous coronary intervention (PCI). The primary endpoint of the OPTIMA-3 is a composite of cardiovascular death, myocardial infarction, ischemic stroke, systemic thromboembolism and unplanned revascularization up to 12 months; the major secondary endpoint is the International Society of Thrombosis and Hemostasis (ISTH) major bleeding or clinically relevant non-major bleeding (CRNMB).

In the OPTIMA-4 sub-study, 1472 subjects who prefer dabigatran will be randomly assigned in a 1:1 ratio to a dual antithrombotic therapy of dabigatran 110 mg twice daily with ticagrelor 90 mg twice daily or with clopidogrel 75 mg od for 12 months after PCI. The primary safety endpoint of the OPTIMA-4 is ISTH major bleeding or CRNMB at 12 months; the primary efficacy endpoint is a composite of cardiovascular death, myocardial infarction, ischemic stroke, systemic thromboembolism and unplanned revascularization.

Other secondary endpoints comprise death (cardiovascular, non- cardiovascular), MI (fatal or non-fatal, Q-wave or non-Q-wave), unplanned revascularization (target or non-target vessel, target or non-target lesion), stent thrombosis (possible, probable, definite), stroke (hemorrhage or ischemic), all bleeding (ISTH and BARC criteria) and net adverse events.

All endpoints will be collected and compared between subgroups and sub-studies during hospitalization and in 1 month (± 7 days), 6 months (± 7 days) and 12 months (± 7 days) for office visits and in 2 weeks (± 7 days), 2 months (± 7 days) and 3 months (± 7 days) for phone call visits.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years;
* ACS patients concomitant non-valvular AF (paroxysmal, persistent and permanent) underwent PCI and new-generation DES implantation;
* CHA2DS2-VASc score ≥ 2;
* Acceptable risk of bleeding at the discretion of the researchers (e.g. HAS-BLED score ≤ 2)
* Consent to participate in the trial

Exclusion Criteria:

* DES implanted in the left main coronary artery
* Cardiogenic shock or Killip III-IV
* STEMI patients with malignant arrhythmias or underwent electrodefibrillation or CPR or with cardiac mechanical complications (heart rupture, ventricular septal perforation, nipple muscle fracture, etc.)
* History of gastrointestinal or intracranial hemorrhage; active bleeding, trauma or major surgery within one month; suspected or diagnosed aortic dissection
* Ischemic stroke with limb dysfunction or dysphasia
* Known allergy or intolerance to the study medications: warfarin, clopidogrel, aspirin, dabigatran, ticagrelor and heparin
* Participating in other ongoing trials
* Planned surgery in 12 months requiring to withdraw the antiplatelet agents
* Planned RFCA or left atrial appendage occlusion in the next 12m
* Abnormal liver or kidney function (ALT ≥ 3 ULN; estimated CrCl < 30 ml/min calculated by Cockcroft-Gault equation); diagnosed liver cirrhosis
* Hematological disease with bleeding tendency; hemoglobin < 100 g/L, platelet count < 100 × 10^9 /L
* Malignancies or life expectancy less than 1 year
* Pregnant (present, suspected, or planned) or lactating woman
* Patients who are taking drugs which may interact with study agents, such as miconazole, ketoconazole, fluconazole, voriconazole, itraconazole, posaconazole, efinaconazole, and rifampicin, etc.
* Patients with any other conditions that may not be suitable to participate in the trial at the discretion of the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3746 (Estimated)
Dates: Start 2018-02-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of OPTIMA-3 | Up to 12 months (± 7 days) after inclusion
  A composite of cardiovascular death, myocardial infarction, ischemic stroke, systemic thromboembolism and unplanned revascularization
Primary safety endpoint of OPTIMA-4 | Up to 12 months (± 7 days) after inclusion
  ISTH major bleeding or CRNMB
Primary efficacy endpoint of OPTIMA-4 | Up to 12 months (± 7 days) after inclusion
  A composite of cardiovascular death, myocardial infarction, ischemic stroke, systemic thromboembolism and unplanned revascularization

SECONDARY OUTCOMES:
Major secondary endpoint of OPTIMA-3 | Up to 12 months (± 7 days) after inclusion
  Major bleeding or clinically relevant non-major bleeding assessed by the ISTH definition
Other secondary endpoints of OPTIMA-3/4 | Up to 12 months (± 7 days) after inclusion
  Death (cardiovascular, non- cardiovascular), MI (fatal or non-fatal, Q-wave or non-Q-wave), unplanned revascularization (target or non-target vessel, target or non-target lesion), stent thrombosis (possible, probable, definite), stroke (hemorrhage or ischemic), all bleeding (ISTH and BARC criteria) and net adverse events

OTHER OUTCOMES:
Adenosine diphosphate (ADP, final concentration 5 μmol/L) induced platelet aggregation (PLADP) | The venous blood will be collected at 7:30 a.m. on the day of discharge and tested within 2 hours.
  The PLADP will be detected by light transmission aggregometry (LTA) to reflect platelet function under the treatment of clopidogrel or ticagrelor.
Arachidonic acid (AA, final concentration 1 mmol/L) induced platelet aggregation (PLAA) | The venous blood will be collected at 7:30 a.m. on the day of discharge and tested within 2 hours.
  The PLAA will be detected by light transmission aggregometry (LTA) to reflect platelet function under the treatment of aspirin.
Trough concentration of dabigatran (Cmin) | The venous blood will be collected at 0.5 hour before dosing after the patients taking at least 3 days of dabigatran and detected after stored below -80℃ for at most 2 months.
  The trough concentration of dabigatran (Cmin) of dabigatran is to be detected by high-performance liquid chromatography-tandem mass spectrometry (HPLC-MS) in OPTIMA-4 trial.
Single nucleotide polymorphisms (SNPs) | The venous blood will be collected at any time during hospitalization and detected after stored below -80℃ for at most 5 years.
  The single nucleotide polymorphisms (SNPs) related to the antithrombotic agents used in different groups will be detected as follows: (1) clopidogrel-related SNPs: CYP2C19 (rs12248560, rs28399504, rs41291556, rs4244285, rs4986893, rs5633701, rs72552267, rs72558186); (2) ticagrelor-related SNPs: SLCO1B1 (rs113681054), OATP1B1 (rs4149056), CYP3A4 (rs62471956, rs56324128), UGT2B7 (rs61361928); (3) dabigatran-related SNP: ABCB1 (rs4148738, rs1045642), CES1 (rs8192935).

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No